CLINICAL TRIAL: NCT02571894
Title: Effects of Identifying and Treating Early, Subclinical Cardiotoxicity on the Long-Term Incidence of Clinical Cardiotoxicity in Women With Breast Cancer, A Prospective Randomized Study: The Cardio-Oncology Breast Cancer Study (COBC)
Brief Title: The Cardio-Oncology Breast Cancer Study
Acronym: COBC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Elham Hedayati, M.D., Ph.D. Senior Consultant, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COBC
Record Dates: First submitted 2015-09-20; First posted 2015-10-08 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Cardiotoxicity; Cardiomyopathies; Breast Cancer
MeSH Terms: conditions — Cardiotoxicity; Cardiomyopathies; Breast Neoplasms | interventions — Therapeutics; Restraint, Physical; epicatechin gallate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observational arm (No Intervention): Participants randomized to observational arm will receive standard oncological followup and care.
- Intervention arm (Experimental): Intervention arm receives standard oncological followup and care + subclinical cardiotoxicity surveillance and treatment.
  Interventions: Other: Subclinical cardiotoxicity surveillance and treatment

INTERVENTIONS:
Other: Subclinical cardiotoxicity surveillance and treatment — Intervention arm receives cardiology assessment and intervention.
  Other Names: Assessment and intervention of cardiac risk factors.; Assessment of biomarkers, echocardiography and ECG.
  Arms: Intervention arm

SUMMARY:
The main objective of this randomized controlled trial is to test the association between standard cardiac risk factors, biomarkers and parameters of echocardiography, electrocardiography, and cardiac magnetic resonance imaging, (predictors) and subsequent occurrence, frequency and severity of clinical or subclinical cardiotoxicity (outcome) within and between-groups, before start of chemotherapy, during treatment and at 1, 5, and 10 years after the completion of the chemotherapy among women with early breast cancer.

DETAILED DESCRIPTION:
Rationale for the study:

Breast cancer is the most common cancer among Swedish women, accounting for a third of all cancer cases among females. The breast cancer incidence has increased from 2596 to more than 8000 breast cancer diagnosis 2011. During the past 40 years, the age-adjusted incidence has doubled. Early adjuvant therapy reduces the risk of dying with about 50%. (Early adjuvant therapies; chemotherapy, antibodies, endocrine therapy, and radiotherapy). Treatment advances have improved survival rates, but treatment-related cardiotoxicity (CT) remains a substantial problem.

In general, earlier treatment of cardiotoxicity offers the best chances of preventing or ameliorating clinical cardiotoxicity. Risk factors should be modified or reduced by treating elevated blood pressure, normalizing lipids, encouraging weight reduction and smoking cessation. Patient-tailored therapy is now possible, especially given the availability of different chemotherapy regimens, safer anthracycline analogs such as liposomal doxorubicin, and cardioprotective medications such as angiotensin converting enzyme (ACE)-inhibitors, angiotensin receptor blockers, and b-blockers. It is now suggested that new cardiac biomarkers and ultrasound techniques can detect cardiotoxicity in its early, subclinical, stages. The investigators hypothesized that biomarkers can be used to detect subclinical cardiotoxicity and that detecting early signs of cardiotoxicity might reduce the number, time-to-onset, and severity of cardiotoxic events.

In present proposal the investigators aim in a randomized study to compare primary cardiac preventive measurements versus standard care.

Objectives of the trial:

1. Primary objective In a randomized study to investigate the cumulative incidence of cardiotoxic events, per randomized arm, before start of chemotherapy, during treatment and at 1, 5, and 10 years after the completion of the chemotherapy.
2. Secondary Objectives To compare the number, time-to-onset, and severity of cardiotoxic events in an experimental group assessed and treated for subclinical cardiotoxicity before start of chemotherapy, during treatment and at 1, 5, and 10 years after the completion of the chemotherapy and a control group receiving standard of care without early assessment for subclinical cardiotoxicity. Data on the same variables will be collected from both groups before start of chemotherapy, during treatment and at 1, 5, and 10 years. Data from the experimental group will be used in real time to guide therapy, but data from the control group will be not be analyzed until after the end of the study.

To assess subclinical cardiotoxicity with serum concentrations of biomarkers, tissue Doppler and strain echocardiography, electrocardiography, and magnetic resonance imaging, as well as with standard cardiac risk assessment based on standard risk factors: a history of heart disease, increasing age, obesity, hypertension, diabetes mellitus, hypercholesterolemia, smoking, parasternal radiotherapy, and the cumulative dose of anthracyclines and trastuzumab.

To assess the association between primary treatment of existing standard cardiac risk factors, biomarkers and parameters of echocardiography, electrocardiography, and cardiac magnetic resonance imaging, (predictors) and subsequent occurrence of clinical or subclinical cardiotoxicity of cardiotoxicity (outcome) within and between-groups, over time.

To examine how a diagnosis of breast cancer and the development of cardiotoxicity influences women's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women with newly diagnosed breast cancer who are eligible to receive neo-adjuvant or adjuvant chemotherapy, with or without trastuzumab, according to the guidelines for breast cancer.
* Written informed consent must be given.

Exclusion Criteria:

* A history of heart disease; ischemic heart disease, arrhythmias, heart failure, and valve diseases.
* Previously received oncological treatment for any malignancy.
* Other disease or conditions that complicates or precludes the patient from following the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 1 year after the completion of the chemotherapy.
  The cumulative incidence of clinical or subclinical cardiotoxicity, per randomized arm, in women with breast cancer at 1 year after treatment with neo- or adjuvant chemotherapy.

SECONDARY OUTCOMES:
Event free survival | 5 and 10 years after the completion of the chemotherapy.
Overall survival | 1, 5 and 10 years after the completion of the chemotherapy.
The levels of serum biomarkers (hs-Troponin T (hs-TnT), B-type natriuretic peptide (BNP)). | 1, 5 and 10 years after the completion of the chemotherapy.
Echocardiographic global longitudinal strain | 1, 5 and 10 years after the completion of the chemotherapy.
The quality of life | 1, 5 and 10 years after the completion of the chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Elham Hedayati, MD, PhD, Principal Investigator — Karolinska University Hospital; Laila Hubbert, MD, PhD, Principal Investigator — University Hospital, Linkoeping
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Autier P, Boniol M, La Vecchia C, Vatten L, Gavin A, Hery C, Heanue M. Disparities in breast cancer mortality trends between 30 European countries: retrospective trend analysis of WHO mortality database. BMJ. 2010 Aug 11;341:c3620. doi: 10.1136/bmj.c3620. PMID 20702548
- [Background] von Minckwitz G, Blohmer JU, Costa SD, Denkert C, Eidtmann H, Eiermann W, Gerber B, Hanusch C, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Kummel S, Paepke S, Schneeweiss A, Untch M, Zahm DM, Mehta K, Loibl S. Response-guided neoadjuvant chemotherapy for breast cancer. J Clin Oncol. 2013 Oct 10;31(29):3623-30. doi: 10.1200/JCO.2012.45.0940. Epub 2013 Sep 3. PMID 24002511
- [Background] Goldhirsch A, Gelber RD, Piccart-Gebhart MJ, de Azambuja E, Procter M, Suter TM, Jackisch C, Cameron D, Weber HA, Heinzmann D, Dal Lago L, McFadden E, Dowsett M, Untch M, Gianni L, Bell R, Kohne CH, Vindevoghel A, Andersson M, Brunt AM, Otero-Reyes D, Song S, Smith I, Leyland-Jones B, Baselga J; Herceptin Adjuvant (HERA) Trial Study Team. 2 years versus 1 year of adjuvant trastuzumab for HER2-positive breast cancer (HERA): an open-label, randomised controlled trial. Lancet. 2013 Sep 21;382(9897):1021-8. doi: 10.1016/S0140-6736(13)61094-6. Epub 2013 Jul 18. PMID 23871490
- [Background] Slamon DJ, Leyland-Jones B, Shak S, Fuchs H, Paton V, Bajamonde A, Fleming T, Eiermann W, Wolter J, Pegram M, Baselga J, Norton L. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med. 2001 Mar 15;344(11):783-92. doi: 10.1056/NEJM200103153441101. PMID 11248153
- [Background] Suter TM, Procter M, van Veldhuisen DJ, Muscholl M, Bergh J, Carlomagno C, Perren T, Passalacqua R, Bighin C, Klijn JG, Ageev FT, Hitre E, Groetz J, Iwata H, Knap M, Gnant M, Muehlbauer S, Spence A, Gelber RD, Piccart-Gebhart MJ. Trastuzumab-associated cardiac adverse effects in the herceptin adjuvant trial. J Clin Oncol. 2007 Sep 1;25(25):3859-65. doi: 10.1200/JCO.2006.09.1611. Epub 2007 Jul 23. PMID 17646669
- [Background] Verma S, Ewer MS. Is cardiotoxicity being adequately assessed in current trials of cytotoxic and targeted agents in breast cancer? Ann Oncol. 2011 May;22(5):1011-1018. doi: 10.1093/annonc/mdq607. Epub 2010 Nov 22. PMID 21097988
- [Background] Ewer MS, Swain SM, Cardinale D, Fadol A, Suter TM. Cardiac dysfunction after cancer treatment. Tex Heart Inst J. 2011;38(3):248-52. PMID 21720462
- [Background] Harbeck N, Ewer MS, De Laurentiis M, Suter TM, Ewer SM. Cardiovascular complications of conventional and targeted adjuvant breast cancer therapy. Ann Oncol. 2011 Jun;22(6):1250-1258. doi: 10.1093/annonc/mdq543. Epub 2010 Nov 26. PMID 21112929
- [Background] Yeh ET, Bickford CL. Cardiovascular complications of cancer therapy: incidence, pathogenesis, diagnosis, and management. J Am Coll Cardiol. 2009 Jun 16;53(24):2231-47. doi: 10.1016/j.jacc.2009.02.050. PMID 19520246
- [Background] Albini A, Pennesi G, Donatelli F, Cammarota R, De Flora S, Noonan DM. Cardiotoxicity of anticancer drugs: the need for cardio-oncology and cardio-oncological prevention. J Natl Cancer Inst. 2010 Jan 6;102(1):14-25. doi: 10.1093/jnci/djp440. Epub 2009 Dec 10. PMID 20007921
- [Background] Perez EA, Suman VJ, Davidson NE, Sledge GW, Kaufman PA, Hudis CA, Martino S, Gralow JR, Dakhil SR, Ingle JN, Winer EP, Gelmon KA, Gersh BJ, Jaffe AS, Rodeheffer RJ. Cardiac safety analysis of doxorubicin and cyclophosphamide followed by paclitaxel with or without trastuzumab in the North Central Cancer Treatment Group N9831 adjuvant breast cancer trial. J Clin Oncol. 2008 Mar 10;26(8):1231-8. doi: 10.1200/JCO.2007.13.5467. Epub 2008 Feb 4. PMID 18250349
- [Background] Nilsson G, Holmberg L, Garmo H, Duvernoy O, Sjogren I, Lagerqvist B, Blomqvist C. Distribution of coronary artery stenosis after radiation for breast cancer. J Clin Oncol. 2012 Feb 1;30(4):380-6. doi: 10.1200/JCO.2011.34.5900. Epub 2011 Dec 27. PMID 22203772
- [Background] Dandel M, Lehmkuhl H, Knosalla C, Suramelashvili N, Hetzer R. Strain and strain rate imaging by echocardiography - basic concepts and clinical applicability. Curr Cardiol Rev. 2009 May;5(2):133-48. doi: 10.2174/157340309788166642. PMID 20436854
- [Background] Fallah-Rad N, Walker JR, Wassef A, Lytwyn M, Bohonis S, Fang T, Tian G, Kirkpatrick ID, Singal PK, Krahn M, Grenier D, Jassal DS. The utility of cardiac biomarkers, tissue velocity and strain imaging, and cardiac magnetic resonance imaging in predicting early left ventricular dysfunction in patients with human epidermal growth factor receptor II-positive breast cancer treated with adjuvant trastuzumab therapy. J Am Coll Cardiol. 2011 May 31;57(22):2263-70. doi: 10.1016/j.jacc.2010.11.063. PMID 21616287
- [Background] Lawley C, Wainwright C, Segelov E, Lynch J, Beith J, McCrohon J. Pilot study evaluating the role of cardiac magnetic resonance imaging in monitoring adjuvant trastuzumab therapy for breast cancer. Asia Pac J Clin Oncol. 2012 Mar;8(1):95-100. doi: 10.1111/j.1743-7563.2011.01462.x. Epub 2012 Jan 12. PMID 22369450
- [Background] Oberholzer K, Kunz RP, Dittrich M, Thelen M. [Anthracycline-induced cardiotoxicity: cardiac MRI after treatment for childhood cancer]. Rofo. 2004 Sep;176(9):1245-50. doi: 10.1055/s-2004-813416. German. PMID 15346258
- [Background] Garrone O, Crosetto N, Lo Nigro C, Catzeddu T, Vivenza D, Monteverde M, Merlano M, Feola M. Prediction of anthracycline cardiotoxicity after chemotherapy by biomarkers kinetic analysis. Cardiovasc Toxicol. 2012 Jun;12(2):135-42. doi: 10.1007/s12012-011-9149-4. PMID 22189487
- [Background] Sawaya H, Sebag IA, Plana JC, Januzzi JL, Ky B, Tan TC, Cohen V, Banchs J, Carver JR, Wiegers SE, Martin RP, Picard MH, Gerszten RE, Halpern EF, Passeri J, Kuter I, Scherrer-Crosbie M. Assessment of echocardiography and biomarkers for the extended prediction of cardiotoxicity in patients treated with anthracyclines, taxanes, and trastuzumab. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):596-603. doi: 10.1161/CIRCIMAGING.112.973321. Epub 2012 Jun 28. PMID 22744937
- [Background] Ky B, Putt M, Sawaya H, French B, Januzzi JL Jr, Sebag IA, Plana JC, Cohen V, Banchs J, Carver JR, Wiegers SE, Martin RP, Picard MH, Gerszten RE, Halpern EF, Passeri J, Kuter I, Scherrer-Crosbie M. Early increases in multiple biomarkers predict subsequent cardiotoxicity in patients with breast cancer treated with doxorubicin, taxanes, and trastuzumab. J Am Coll Cardiol. 2014 Mar 4;63(8):809-16. doi: 10.1016/j.jacc.2013.10.061. Epub 2013 Nov 27. PMID 24291281
- [Background] Alehagen U, Dahlstrom U, Rehfeld JF, Goetze JP. Prognostic assessment of elderly patients with symptoms of heart failure by combining high-sensitivity troponin T and N-terminal pro-B-type natriuretic peptide measurements. Clin Chem. 2010 Nov;56(11):1718-24. doi: 10.1373/clinchem.2009.141341. Epub 2010 Sep 15. PMID 20844063
- [Background] Maisel A, Mueller C, Nowak R, Peacock WF, Landsberg JW, Ponikowski P, Mockel M, Hogan C, Wu AH, Richards M, Clopton P, Filippatos GS, Di Somma S, Anand I, Ng L, Daniels LB, Neath SX, Christenson R, Potocki M, McCord J, Terracciano G, Kremastinos D, Hartmann O, von Haehling S, Bergmann A, Morgenthaler NG, Anker SD. Mid-region pro-hormone markers for diagnosis and prognosis in acute dyspnea: results from the BACH (Biomarkers in Acute Heart Failure) trial. J Am Coll Cardiol. 2010 May 11;55(19):2062-76. doi: 10.1016/j.jacc.2010.02.025. PMID 20447528
- [Background] Alehagen U, Dahlstrom U, Rehfeld JF, Goetze JP. Association of copeptin and N-terminal proBNP concentrations with risk of cardiovascular death in older patients with symptoms of heart failure. JAMA. 2011 May 25;305(20):2088-95. doi: 10.1001/jama.2011.666. PMID 21610241
- [Background] Goetze JP, Alehagen U, Flyvbjerg A, Rehfeld JF. Making sense of chromogranin A in heart disease. Lancet Diabetes Endocrinol. 2013 Sep;1(1):7-8. doi: 10.1016/S2213-8587(13)70035-4. Epub 2013 Jun 13. No abstract available. PMID 24622255
- [Background] Chisalita SI, Dahlstrom U, Arnqvist HJ, Alehagen U. Increased IGF1 levels in relation to heart failure and cardiovascular mortality in an elderly population: impact of ACE inhibitors. Eur J Endocrinol. 2011 Dec;165(6):891-8. doi: 10.1530/EJE-11-0584. Epub 2011 Oct 5. PMID 21976623
- [Background] Crone SA, Zhao YY, Fan L, Gu Y, Minamisawa S, Liu Y, Peterson KL, Chen J, Kahn R, Condorelli G, Ross J Jr, Chien KR, Lee KF. ErbB2 is essential in the prevention of dilated cardiomyopathy. Nat Med. 2002 May;8(5):459-65. doi: 10.1038/nm0502-459. PMID 11984589
- [Background] Bozkurt B, Mann DL, Deswal A. Biomarkers of inflammation in heart failure. Heart Fail Rev. 2010 Jul;15(4):331-41. doi: 10.1007/s10741-009-9140-3. PMID 19363700
- [Background] Rumsfeld JS, Alexander KP, Goff DC Jr, Graham MM, Ho PM, Masoudi FA, Moser DK, Roger VL, Slaughter MS, Smolderen KG, Spertus JA, Sullivan MD, Treat-Jacobson D, Zerwic JJ; American Heart Association Council on Quality of Care and Outcomes Research, Council on Cardiovascular and Stroke Nursing, Council on Epidemiology and Prevention, Council on Peripheral Vascular Disease, and Stroke Council. Cardiovascular health: the importance of measuring patient-reported health status: a scientific statement from the American Heart Association. Circulation. 2013 Jun 4;127(22):2233-49. doi: 10.1161/CIR.0b013e3182949a2e. Epub 2013 May 6. No abstract available. PMID 23648778
- [Background] Rector TS, Cohn JN. Assessment of patient outcome with the Minnesota Living with Heart Failure questionnaire: reliability and validity during a randomized, double-blind, placebo-controlled trial of pimobendan. Pimobendan Multicenter Research Group. Am Heart J. 1992 Oct;124(4):1017-25. doi: 10.1016/0002-8703(92)90986-6. PMID 1529875
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Sprangers MA, Groenvold M, Arraras JI, Franklin J, te Velde A, Muller M, Franzini L, Williams A, de Haes HC, Hopwood P, Cull A, Aaronson NK. The European Organization for Research and Treatment of Cancer breast cancer-specific quality-of-life questionnaire module: first results from a three-country field study. J Clin Oncol. 1996 Oct;14(10):2756-68. doi: 10.1200/JCO.1996.14.10.2756. PMID 8874337
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. J Gen Intern Med. 2007 Nov;22(11):1596-602. doi: 10.1007/s11606-007-0333-y. Epub 2007 Sep 14. PMID 17874169
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Peto R, Davies C, Godwin J, Gray R, Pan HC, Clarke M, Cutter D, Darby S, McGale P, Taylor C, Wang YC, Bergh J, Di Leo A, Albain K, Swain S, Piccart M, Pritchard K. Comparisons between different polychemotherapy regimens for early breast cancer: meta-analyses of long-term outcome among 100,000 women in 123 randomised trials. Lancet. 2012 Feb 4;379(9814):432-44. doi: 10.1016/S0140-6736(11)61625-5. Epub 2011 Dec 5. PMID 22152853
- [Background] EBCTCG (Early Breast Cancer Trialists' Collaborative Group); McGale P, Taylor C, Correa C, Cutter D, Duane F, Ewertz M, Gray R, Mannu G, Peto R, Whelan T, Wang Y, Wang Z, Darby S. Effect of radiotherapy after mastectomy and axillary surgery on 10-year recurrence and 20-year breast cancer mortality: meta-analysis of individual patient data for 8135 women in 22 randomised trials. Lancet. 2014 Jun 21;383(9935):2127-35. doi: 10.1016/S0140-6736(14)60488-8. Epub 2014 Mar 19. PMID 24656685
- [Background] Tarantini L, Cioffi G, Gori S, Tuccia F, Boccardi L, Bovelli D, Lestuzzi C, Maurea N, Oliva S, Russo G, Faggiano P; Italian Cardio-Oncologic Network. Trastuzumab adjuvant chemotherapy and cardiotoxicity in real-world women with breast cancer. J Card Fail. 2012 Feb;18(2):113-9. doi: 10.1016/j.cardfail.2011.10.015. Epub 2011 Dec 3. PMID 22300778
- [Background] Dinse GE, Lagakos SW. Nonparametric estimation of lifetime and disease onset distributions from incomplete observations. Biometrics. 1982 Dec;38(4):921-32. PMID 7168795
- [Background] Smith DP. Regression analysis of "current status" life tables on duration of breastfeeding in Sri Lanka. Soc Biol. 1985 Spring-Summer;32(1-2):90-101. doi: 10.1080/19485565.1985.9988595. PMID 4081811